CLINICAL TRIAL: NCT05654064
Title: Comparison of Remifentanil-dexmedetomidine and Dexmedetomidine-fentanyl Sedation Protocols for Pregnant Patients Undergoing Minimally Invasive Fetoscopic Procedures
Brief Title: Comparing Fetoscopic Surgery Protocols
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Deferred by IRB.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022-0168
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Minimally Invasive Fetoscopic Procedures

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participant and surgeon will be blinded to which combination of medications are used during the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remifentanil-dexmedetomidine (Active Comparator)
  Interventions: Drug: Remifentanil-dexmedetomidine
- Dexmedetomidine- fentanyl (Active Comparator)
  Interventions: Drug: Dexmedetomidine-fentanyl

INTERVENTIONS:
Drug: Remifentanil-dexmedetomidine — Compare adequacy of remifentanil-dexmedetomidine sedation protocols in pregnant patients undergoing minimally invasive fetoscopic procedures.
  Arms: Remifentanil-dexmedetomidine
Drug: Dexmedetomidine-fentanyl — Compare adequacy of dexmedetomidine-fentanyl sedation protocols in pregnant patients undergoing minimally invasive fetoscopic procedures.
  Arms: Dexmedetomidine- fentanyl

SUMMARY:
Determine surgeon and patient satisfaction with remifentanil-dexmedetomidine (REMI) and dexmedetomidine-fentanyl (DEX) sedation protocols in pregnant patients undergoing minimally invasive fetoscopic procedures

ELIGIBILITY:
Inclusion Criteria:

Pregnant patients undergoing one of the following procedures

* Laser photocoagulation of abnormal anastomotic vessels in patients with a twin-twin transfusion syndrome
* Selective radiofrequency ablation or fetoscopic cord coagulation in patients with TRAP sequence or in the presence of intrauterine death of one twin
* Vesicoamniotic shunts or placement of amnioports in patients with LUTO
* Placement of amnioports in patients with oligohydramnios or anhydramnios
* Fetal thoracentesis or placement of thoracoamniotic shunts in patients with congenital pulmonary airway malformation or fetal hydrothorax
* FETO (fetoscopic endotracheal occlusion) as well as balloon removal in patients with congenital diaphragmatic hernia and laser release of amniotic bands

Exclusion Criteria:

Pregnant patients undergoing fetoscopic procedures requiring the following

* Additional procedures (e.g. cerclage)
* Laparotomy with uterine exteriorization to access the uterine cavity
* General anesthesia
* Mid-gestation neural tube defect repair
* EXIT procedures
* Preoperative opioid use
* Diagnosed substance abuse
* Moderate to severe obstructive sleep apnea
* History of allergic reactions to medications to be administered during the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant females undergoing fetoscopic procedures
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Determine surgeon satisfaction with remifentanil-dexmedetomidine sedation | Immediately after procedure completion
  Surgeons will use a scale of 1-4, 1 - Excellent, 2 - Good, 3 - Moderate, 4 - Inadequate
Determine surgeon satisfaction with dexmedetomidine-fentanyl sedation | Immediately after procedure completion
  Surgeons will use a scale of 1-4, 1 - Excellent, 2 - Good, 3 - Moderate, 4 - Inadequate
Determine patient satisfaction with remifentanil-dexmedetomidine sedation | 6 hours after procedure completion
  Iowa Satisfaction with Anesthesia Scale (ISAS) 11 question survey rating anesthesia experience. Six response options from disagree very much to agree very much
Determine patient satisfaction with dexmedetomidine-fentanyl sedation | 6 hours after procedure completion
  Iowa Satisfaction with Anesthesia Scale (ISAS) 11 question survey rating anesthesia experience. Six response options from disagree very much to agree very much

SECONDARY OUTCOMES:
Sedation scores | Every 15 minutes from start of procedure to one hour post-operative
  Assessment of sedation level using a 1 - 5 scale; 1 - No response after name is called loudly with mild shaking, 2 - Responds only after name called loudly and after mild shaking of the body, 3 - Responds only after name called loudly or repeatedly, 4 - Lethargic response to name spoken in normal tone, 5 - Awake and responds to name spoken in normal tone
Side-effect measures | Up 24 hours after procedure
  Incidences of medication side effects will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Mario Patino, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati